CLINICAL TRIAL: NCT03904758
Title: Extraesophageal Reflux - Feasibility of Measurement of Pepsin in Saliva as a Diagnostic Option
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-ENT-Pepsin
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Extraesophageal Reflux
Keywords: extraesophageal reflux; laryngopharyngeal reflux; pepsin; saliva; oropharyngeal pH monitoring; esophageal impedance
MeSH Terms: conditions — Laryngopharyngeal Reflux

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into two study arms.
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitoring of pH with Restech (Experimental): The patients with EER randomized into this arm will undergo pH monitoring using Restech system
  Interventions: Diagnostic Test: Pepsin in saliva test
- Monitoring of oesophageal impedance (Experimental): The patients with EER randomized into this arm will undergo monitoring of oesophageal impedance
  Interventions: Diagnostic Test: Pepsin in saliva test

INTERVENTIONS:
Diagnostic Test: Pepsin in saliva test — The presence of pepsin in the saliva will be tested in both groups of patients.

SUMMARY:
The diagnostics of extraesophageal reflux (EER) is challenging. Currently, 24-h dual-probe esophageal pH monitoring or impedance is considered the best diagnostic method for EER. The 24-h oropharyngeal pH monitoring is a newer method aimed at detecting episodes of reflux to the oropharynx. Unfortunately, all these methods have many disadvantages. Pepsin detection in saliva would be an almost ideal diagnostic technique. However, data of its reliability is lacking. The aim of the study is to compare results of oropharyngeal pH monitoring and esophageal impedance monitoring, compared to a quantified pepsin presence in the saliva obtained immediately prior to 24-hour monitoring and to evaluate the feasibility of this technique as a routine option of diagnosing the presence of extraesophageal reflux.

DETAILED DESCRIPTION:
Extraesophageal reflux (EER) has recently been found to be a risk factor for many head and neck pathologies. Many studies have shown that contact between the refluxed content and mucous tissue can cause local inflammation and edema and thus facilitate the development of inflammation. Although important, the diagnostics of EER is not easy. The simplest means of collecting information about reflux problems is questioning potential sufferers. However, although many questionnaires have been developed over the last few years, questioning is still not a suitable technique for the evaluation of EER, the reason being that symptoms of EER are heterogeneous and very common. Currently, 24-h dual-probe esophageal pH monitoring or impedance is considered the best diagnostic method for EER. The 24-h oropharyngeal pH monitoring is a newer method aimed at detecting episodes of reflux to the oropharynx and seems to generate similar results. However, these methods may not be tolerated well. Moreover, the position of the sensor, which is placed in the hypopharynx or oropharynx, does not precisely reflect the amount of reflux content that reaches larynx, nasopharynx, nasal cavity or middle ear. Another disadvantage of pH monitoring is that it enables only a short-term analysis over a timespan of just 24-48 h. Detection of pepsin in fluids and tissues is considered by some authors to be perhaps more appropriate than pH monitoring because it reflects the long-term effects of EER and proves that EER is truly affecting the examined region. This is particularly true for more distant regions like the middle ear. Pepsin detection in saliva would be very well tolerated and fast diagnostic method. However, data of its reliability are lacking. The aim of the study is to compare results of oropharyngeal pH monitoring and esophageal impedance monitoring, compared to a quantified pepsin presence in the saliva obtained immediately prior to 24-hour monitoring and to evaluate the feasibility of this diagnostic option as a routine method.

ELIGIBILITY:
Inclusion Criteria:

- suspicion of EER indicated for diagnostics

Exclusion Criteria:

* head and neck cancer
* not-signing of the informed consent with participation in the study
* intolerance of 24-hour monitoring
* treatment with proton pump inhibitors

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Reflux symptom index (RSI) | 24 hours
  Reflux symptom index is a standard tool in the form of a questionnaire scale where the patients evaluate their problems related to reflux on a scale of 0 (no problems) to 5 (severe). The value of RSI over 13 may be indicative of serious reflux-related problems.
Reflux finding score (RFS) | 24 hours
  Reflux finding score is a standard tool for assessing the presence and severity of reflex, evaluating reflux symptoms in eight areas.

SECONDARY OUTCOMES:
Presence of pepsin in the saliva | 24 hours
  The presence of pepsin in the saliva will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Formánek, MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data with other researchers.